CLINICAL TRIAL: NCT04452422
Title: High Prevalence of Deep Venous Thrombosis in Non-severe COVID-19 Patients Hospitalized for a Neurovascular Pathology
Brief Title: Deep Venous Thrombosis in Non-severe COVID-19 Patients Hospitalized for a Neurovascular Pathology
Acronym: VT-Covid-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7908
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2020-06

CONDITIONS: Deep Venous Thrombosis
Keywords: non-severe COVID-19; neurovascular diseases; Doppler ultrasound; Deep venous thrombosis; Covid-19; SARS-CoV-2
MeSH Terms: conditions — Venous Thrombosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe SARS-CoV-2 infection, responsible of COVID-19, is accompanied by many venous thromboembolic events. Antithrombotic treatment is the cornerstone of management of many neurovascular diseases (NVDs) and the benefit-risk ratio is crucial to avoid hemorrhagic complications. Therefore, in non-severe COVID-19 patients affected by NVDs, the diagnostic of deep venous thrombosis (DVT) is challenging. Using bedside Doppler ultrasonography (DUS) of lower limbs, this study investigated the rates of DVT in these patients in stroke unit.

ELIGIBILITY:
* Inclusion criteria:

  * Age>18 years
  * COVID-19 confirmed with RT-PCER and/or chest CT-scan
  * Acute neurovascular disease defined as transient ischemic attack or acute ischemic stroke or venous cerebral thrombosis or hemorrhagic stroke.
* Exclusion criteria:

  * age<18
  * Other neurovascular diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with COVID-19 confirmed with RT-PCER and/or chest CT-scan and with acute neurovascular disease defined as transient ischemic attack or acute ischemic stroke or venous cerebral thrombosis or hemorrhagic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Number of cumulated deep venous thrombosis among the hospitalization | Day 7 after admisssion

CONTACTS AND LOCATIONS:
Locations (1):
- Service Unité Neurovasculaire, Strasbourg, France